CLINICAL TRIAL: NCT00875914
Title: Randomized Comparison Between Magnetically Navigated vs Manually Guided Radiofrequency in AV-node-reentry-tachycardia
Brief Title: Magnetically Navigated vs. Manually Guided Radiofrequency in Atrioventricular-node-reentry-tachycardia
Acronym: MAGMA-AVNRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Gabi Hessling MD, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. C00909
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Atrioventricular Nodal Reentry Tachycardia; Radiofrequency Ablation
Keywords: AV-node reentry tachycardia; radiofrequency ablation; magnetic navigation system
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manually guided (Experimental): Treatment with manually guided RF-catheter
  Interventions: Procedure: RF-ablation
- Magnetically navigated (Experimental): Treatment with magnetically navigated RF-catheter.
  Interventions: Procedure: RF-ablation

INTERVENTIONS:
Procedure: RF-ablation — 4mm-tip catheter manually guided vs magneticallly navigated

SUMMARY:
The MAGMA-AVNRT study compares two different methods of handling the ablation catheters for av-node-reentry-tachycardia with regard to x-ray dose, safety and success: manually guided vs magnetically navigated RF-catheter.

DETAILED DESCRIPTION:
AV-node reentry tachycardia can be treated by radiofrequency ablation or modulation of the slow pathway of the av node. The success rate is 90 to 95%.

There are different options to navigate the ablation catheter: manually guided vs magnetically guided.

For magnetic guidance two magnets are positioned beneath the patient. A mangetic field is induced and a catheter with a ferromagnetic tip can be navigated from outside with a joystick by modifying the vectors of the magnetic field.

We hypothesized that a magnetic guidance of the RF-ablation catheter results in lower x-ray time and dose for the patient and the physician with comparable safety und success rates.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* suspected AV-node-reentry-tachycardia
* written informed consent

Exclusion Criteria:

* pregnancy
* contraindication against electrophysiological study or ablation
* congenital heart disease or other anatomical abnormalities
* previous surgical procedure involving atrium except aorto-coronary bypass grafts
* psychiatric disease that makes a completion of study improbable
* severe comorbidities with a life expectancy less than 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Total x-ray time and dose for patient | electrophysiological examination

SECONDARY OUTCOMES:
X-ray time and dose for physician | electrophysiological study
Safety of ablation (AV-Block, perforation) | end of electrophysiological study
short-term and long-term-success | end of procedure and 6 months after procedure
number of RF-application | procedure
Duration of electrophysiological study (ablation included) | procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Hessling, MD, Study Chair — Deutsches Herzzentrum München; Peter Schuster, MD, Study Chair — University of Bergen; Isabel Deisenhofer, MD, Study Chair — Deutsches Herzzentrum München
Locations (1):
- University Hospital Bergen, Bergen, Norway